CLINICAL TRIAL: NCT03333577
Title: Evaluation of the Baha SoundArc in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM5714
Record Dates: First submitted 2017-11-02; First posted 2017-11-07 (Actual); Results first posted 2019-04-11 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Hearing Loss, Conductive; Hearing Loss, Mixed; Hearing Loss, Unilateral
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Hearing Loss, Unilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experimental SoundArc study group (Experimental): all subjects will receive the SoundArc intervention
  Interventions: Device: SoundArc

INTERVENTIONS:
Device: SoundArc — non-surgical attachment method for wearing a bone conduction hearing system

SUMMARY:
The purpose of this study is to gather clinical performance data on the Baha SoundArc

DETAILED DESCRIPTION:
Current Baha recipients that are using a Baha SoftBand will be recruited to be fitted with an alternative non-surgical option for using their Baha Sound Processor. The subjects will be tested with there existing Baha Sound Processor on the SoftBand and will then be fitted with the Baha SoundArc where they will perform a one month take home trial. At the end of this trial, the subject will return for testing and evaluation of their experience with this new fitting option.

ELIGIBILITY:
Inclusion Criteria:• Existing recipients using a Baha sound processor on a Softband for at least three months

* Subjects aged 5 through 12 years of age
* Subjects should be able to perform clinical testing adapted for age and developmental status, (Threshold sound field audiometry and basic monosyllabic word test, PBK)
* Willingness on behalf of the subject's parent or guardian to complete study questionnaire

Exclusion Criteria:• Subject's inability to perform requisite test measures as described in the study protocol

-

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Cire, Study Director — Study Director
Locations (3):
- United States (3):
  - Arizona Hearing and Balance, Chandler, Arizona
  - Rady Children's Hospital, San Diego, California
  - Cook Children's Hospital, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moyer C, Purdy J, Carvalho D, Vaughan L, Shroyer L. Evaluation of the Baha SoundArc in children. Int J Pediatr Otorhinolaryngol. 2024 Apr;179:111925. doi: 10.1016/j.ijporl.2024.111925. Epub 2024 Mar 27. PMID 38552429

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental SoundArc Study Group
Started | 32
Completed | 25
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Experimental SoundArc Study Group
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants] — Population: 25 subjects completed visit 1 and 2 and were analyzed
  Participants
    <=18 years | 25
    Between 18 and 65 years | 0
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 25 subjects completed visit 1 and 2 and were analyzed
  Participants
    Female | 9
    Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction Survey
Description: To evaluate patient experience when using the Baha SoundArc after a one month take-home trial, compared to the existing Baha Softband on the Participant Take Home questionnaire (strongly agree, Agree, Neutral, disagree, strongly disagree)
Time Frame: one month post fitting
Measure: Number; unit: percentage of satisfied subjects
Arm/Group | Experimental SoundArc Study Group
Number analyzed (Participants) | 25
percentage of satisfied subjects | 65

2. Primary Outcome: Percentage Correct on Word Identification Task
Description: one list of monosyllabic words (PBK words) was assessed at 60dBA, with word scores recorded as a percent correct.
Time Frame: 4 weeks post fitting
Measure: Mean (Standard Deviation); unit: % corrrect words
Arm/Group | Experimental SoundArc Study Group
Number analyzed (Participants) | 25
% corrrect words | 85.1 (13.6)

ADVERSE EVENTS:
Time Frame: Study duration use one month interval. Adverse events were recorded from time of consent/enrollment until completion of study
Description: Adverse events were recorded from time of consent/enrollment until completion of study
Arm/Group | Experimental SoundArc Study Group
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental SoundArc Study Group (N=25)
irritation from use of Device (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT03333577/Prot_000.pdf